CLINICAL TRIAL: NCT06377137
Title: High Intensity Training Based on Small-sided Soccer Games for Health: Effects on Cardiometabolic Health, Motor Performance and Adherence to 24-hour Movement Guidelines in Adolescents With Overweight and Metabolic Dysfunction
Brief Title: High-intensity Small-sided Soccer Games for Cardiometabolic Health in Adolescents With Metabolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Hélder Fonseca, Assistant Professor, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: University of the Porto
Record Dates: First submitted 2024-04-01; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Adolescent; Metabolic Syndrome
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Small-sided soccer games groups (SSSG) (Experimental): SSSG will perform 16 weeks of training, 3 sessions/week, and ~55 minutes/session. Each session will begin with a 15-minute warm-up, 32 minutes of principal activity, and 5 minutes of cool down. The SSSG will consist of a program based on high-intensity SSSG.
  The training protocol is based on a pilot study conducted to characterize the exertion profile. The SSSG will be performed in a fractional regimen of 8 sets of 4 minutes and 2 minutes rest. The format of the SSGs will be 3v3, although they can be adapted to 2v2 or 4v4 when necessary. In addition, it will take place in a playing area of 9 x 18 meters equivalent to 27 square meters per player. To encourage high intensity, the following will be used (i) man-to-man marking; (ii) to score a goal, the entire team must be in the opponent's half of the field; (iii) balls will be available to reduce stoppages in play; (iv) the coach will motivate the team to maintain high intensity.
  Interventions: Behavioral: Small-sided soccer games groups (SSSG)
- Traditional soccer training groups (TSG) (Experimental): SSSG will perform 16 weeks of training, 3 sessions/week, and ~55 minutes/session. Each session will begin with a 15-minute warm-up, 32 minutes of principal activity, and 5 minutes of cool down.
  The TSG group will base its training on 30 minutes of technical exercises with the ball individually or in pairs (dribbling, shooting and passing), ending with 10 minutes of a match organized according to the original characteristics of an indoor soccer game.
  Interventions: Behavioral: Traditional soccer training groups (TSG)
- Control Group (CG) (No Intervention): CG will perform only regular school physical education classes without any additional intervention

INTERVENTIONS:
Behavioral: Small-sided soccer games groups (SSSG) — Physical exercise intervention
  Arms: Small-sided soccer games groups (SSSG)
Behavioral: Traditional soccer training groups (TSG) — Physical exercise intervention
  Arms: Traditional soccer training groups (TSG)

SUMMARY:
Pediatric obesity is considered one of the most important public health problems worldwide due to its high prevalence and associated comorbidities. Physical exercise has been shown to have an important role in the treatment of obesity and associated cardiometabolic dysfunction. Small-sided soccer games (SSSG) have been explored as a promising way of increasing physical exercise due to its benefits on cardiometabolic health and high degree of enjoyment, which favors long-term adherence.

The objective of this research is to determine the effects of a 16-week high-intensity SSSG-based exercise intervention on cardiometabolic risk factors, physical fitness, adherence to 24-hour movement patterns, enjoyment and adherence to the intervention in adolescents with metabolic dysfunction and compare them to the effects of a traditional soccer intervention.

The investigators hypothesize that high-intensity SSSG are more effective in improving the obesity-related cardiometabolic risk profile in adolescents with cardiometabolic dysfunction compared to traditional soccer training.

A parallel 3-arm randomized controlled trial will be conducted in adolescents with overweight and metabolic dysfunction between 11 and 15 years of age. The inclusion criteria are: (i) age between 11-15 years at the time of intervention start; (ii) overweight or obesity (BMI> 85th percentile); (iii) Abdominal obesity ≥90th percentile as assessed by waist circumference or a waist-to-height ratio ≥ 0.5; (iv) willing to participate in the study regardless of possible group allocation; (v) informed consent given by participant and legal representatives. Exclusion criteria: (i) health condition not compatible with participation in physical exercise; (ii) history of recent musculoskeletal injury hindering exercise participation; (iii) concurrent participation in a structured weight loss or exercise program.

Those eligible to participate in the study will be randomly assigned to one of three groups: i) SSSG group, ii) traditional soccer play group (TSG), or, iii) non-exercise intervention control group (CG). Participants in both exercise intervention groups will undergo a 16-week intervention. The SSSG group will participate in a high-intensity small-sided soccer games training, while the TSG will undergo a technical and tactical skills training program and traditional soccer training. The CG participants will continue with regular school physical education classes without any additional intervention. Before and after the intervention, all participants will be assessed for cardiometabolic and hepatic biochemical markers, physical fitness, anthropometry and body composition, blood pressure, objective daily physical activity and sleep quality, and perceived enjoyment of participation in SSSG and TSG. The primary outcomes of the study will be waist circumference and cardiorespiratory fitness.

The study protocol was approved by the Ethics Committee of the Faculty of Sport of the University of Porto and by the Scientific Ethics Committee of the Adventist University of Chile.

ELIGIBILITY:
Inclusion Criteria:

* Age between 11-15 years at the time of intervention start
* Overweight or obesity (BMI> 85th percentile)
* Abdominal obesity ≥90th percentile as assessed by waist circumference or a waist-to- height ratio ≥ 0.5
* Willing to participate in the study regardless of possible group allocation
* Informed consent given by participant and legal representatives

Exclusion Criteria:

* Health condition not compatible with participation in physical exercise
* History of recent musculoskeletal injury hindering exercise participation
* Concurrent participation in a structured weight loss or exercise program

Ages: 11 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 16 weeks
  Anthropometric measurement of abdominal obesity; cm
Cardiorespiratory fitness | 16 weeks
  1-mile walk/run test; minutes to run 1 mile

SECONDARY OUTCOMES:
Variation in fasting blood glucose concentration (mg/dL) | 16 weeks
  Variation in fasting blood glucose concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in serum insulin concentration (mU/L) | 16 weeks
  Variation in serum insulin concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in HOMA-IR | 16 weeks
  Variation in HOMA-IR after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in glycosylated hemoglobin concentration (mg/dL) | 16 weeks
  Variation in Glycosylated hemoglobin concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in high-density lipoprotein cholesterol concentration (mg/dL) | 16 weeks
  Variation in High-density lipoprotein cholesterol concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in low-density lipoprotein cholesterol concentration (mg/dL) | 16 weeks
  Variation in low-density lipoprotein cholesterol concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in total cholesterol concentration (mg/dL) | 16 weeks
  Variation in total cholesterol concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in blood triglycerides concentration (mg/dL) | 16 weeks
  Variation in blood triglycerides concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in blood Alanine aminotransferase concentration (U/L) | 16 weeks
  Variation in blood Alanine aminotransferase concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in blood Aspartate aminotransferase concentration (U/L) | 16 weeks
  Variation in blood Aspartate aminotransferase concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
Variation in blood Gamma glutamyl transferase concentration (U/L) | 16 weeks
  Variation in blood Gamma glutamyl transferase concentration after 16 weeks of intervention.
  Blood samples will be obtained from each subject early in the morning by venipuncture from the antecubital vein, following a 10-h overnight fast.
6-minute walk test | 16 weeks
  Distance covered walking in 6 minutes.
Hand grip strength | 16 weeks
  Hand grip strength test measured with a digital hand dynamometer
Lower limb strength | 16 weeks
  Assessed by Horizontal jump test.
Body composition | 16 weeks
  Assessed by the electrical bioimpedance method
Body mass index | 16 weeks
  Weight and height will be combined to report BMI in kg/m^2
Neck circumference | 16 weeks
  Assessed by anthropometric techniques
Blood Pressure (mmHg) | 16 weeks
  Systolic and diastolic blood pressure measured with digital sphygmomanometer
Physical activity | 16 weeks
  Physical activity will be assessed objectively with a triaxial accelerometer used 24h/d during 7 consecutive days.
Sleep quality | 16 weeks
  Sleep quality will be assessed objectively with a triaxial accelerometer used 24h/d during 7 consecutive days.
Perceived enjoyment of physical activity | 16 weeks
  Assessed by the Physical Activity Enjoyment Scale questionnaire (PACES). Raw scores are transformed into a scale from 16 to 80. Higher scores correspond to higher perceived enjoyment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No